CLINICAL TRIAL: NCT03289247
Title: A Prospective Single-blinded Randomized Controlled Study Evaluating Efficacy of Tissue Adhaesive in Wound Closure Following Primary Total Knee Arthroplasty
Brief Title: Tissue Adhaesive in Wound Closure Following Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kirill Gromov, MD, PhD, Ass. professor, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HVH-SBTKA-Adhaesive
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Total Knee Arthroplasty; Infection; Arthroplasty Complications
MeSH Terms: conditions — Infections | interventions — Tissue Adhesives

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigator evaluating primary outcome is blinded to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular (No Intervention): Regular closure:
  The standard 3-layer closure is performed using: 1) size 2 coated VICRYL® Plus Antibacterial suture for capsule closure 2) size 2-0 coated VICRYL® Plus Antibacterial suture for subcutaneous tissue closure and 3) stainless steel stables using PROXIMATE® Fixed-Head stapler for cutaneous closure.
- Additional tissue adhaesive (Experimental): The standard 3-layer closure is performed using: 1) size 2 coated VICRYL® Plus Antibacterial suture for capsule closure 2) size 2-0 coated VICRYL® Plus Antibacterial suture for subcutaneous tissue closure and 3) stainless steel stables using PROXIMATE® Fixed-Head stapler for cutaneous closure. tissue adhesive (Leukosan®) is applied on top of the staples according to manufacturer instructions. One layer (one tube) of tissue adhesive is applied following air-drying for 30 seconds, followed by a placement of a second layer with a second layer (one tube), and a second air-drying period of 60 seconds
  Interventions: Device: tissue adhesive (Leukosan®)

INTERVENTIONS:
Device: tissue adhesive (Leukosan®) — Tissue ahaesive
  Arms: Additional tissue adhaesive

SUMMARY:
The study's primary objective is to compare the following parameters between wound closure following primary TKA with and without supplement tissue adhesive (Leukosan®):

DETAILED DESCRIPTION:
Prolonged wound drainage following total joint replacement surgery has been shown to be a predictor of Periprosthetic Joint Infection (PJI) 1-3. Several studies have highlighted this subject, and estimates of the risk of postoperative infection range from 1.3% to 50% among patients with persistent wound drainage 4. Such infections can be one of the most challenging complications following joint replacement surgery and is one of the leading causes of revision surgery following primary hip and knee arthroplasty 5,6.

Several patient-related factors have been associated with delayed wound healing and increased risk of infection following joint replacement surgery. Obesity 4,7, diabetes 8, smoking 9,10 and autoimmune disease 11 have been shown to have a detrimental effect on wound healing. Recently there has also been reports that patients with hypertension 12 have impaired wound healing following total hip arthroplasty (THA) and total knee arthroplasty (TKA).

Surgery related factors such as surgical approach, pneumatic tourniquet time and use of peri-articular local anesthesia have also been shown to have an effect on postoperative wound oozing 9,13.

Finally, several pharmacological factors, such as thromboembolic chemoprophylaxis 4, steroid treatment 9,14 and possibly statins 15,16 might also influence wound healing.

In recent years tissue adhesives for wound closure have been introduced as a replacement or a supplement to conventional closure techniques. Currently very few studies investigate the effect of such tissue adhesives in Total Knee Arthroplasty, and high quality randomized controlled trials (RCT) are lacking.

In this project we wish to:

Evaluate the effect of supplemental wound closure using a high viscosity tissue adhaesive (Leukosan®) in primary TKA with respect to postoperative wound drainage and wound healing.

This project is carried out as a randomized single-blinded controlled trial, in which the clinical outcomes after wound closure following primary bilateral simultaneous TKA with either 1) standard 3-layer closure methods with skin staples or 2) 3-layer closure methods with skin staples supplemented with tissue adhesive (Leukosan®) are compared.

After written informed consent is obtained patients scheduled for a primary bilateral simultaneous TKA will be enrolled in this study and left knee will be randomized to receive either 1) standard 3-layer closure methods with skin staples or 2) 3-layer closure methods with skin staples supplemented with tissue adhesive (Leukosan®), with the opposite treatment on the contralateral knee. All patients will receive AGC total knee prosthesis in both knees (department standard). The standard 3-layer closure consist of: size 2 coated VICRYL® Plus Antibacterial suture for capsule closure, size 2-0 coated VICRYL® Plus Antibacterial suture for subcutaneous tissue closure and stainless steel staples using PROXIMATE® Fixed-Head stapler for cutaneous closure. Wound oozing will be assessed by project nurses during postoperative day 1-3 as well as patient reported wound oozing on postoperative day 3-21. Wound healing will be assessed using ASEPSIS 17,18 score 3 weeks postoperatively.

Range of motion (ROM) will also be recorded at 3 months postoperatively. Allocation of the participants to one of the two treatment groups is done intraoperatively after initial incision has been made. Participants as well as the research coordinator handling the collected questionnaires postoperatively and evaluating wound healing are all unaware of which method was used for skin closure.

Recruitment of participants to this project is expected to begin in September 2015 or as soon as permission from the Regional Ethics Committee and the Danish Data Protections Agency is obtained. A total of 30 participants are to be included at our institution. Recruitment is expected completed after a maximum period of 1.5 years. The project is expected to be completed 1 year after recruitment of the last participant (2018).

ELIGIBILITY:
Inclusion criteria

* Patient > 18 years of age.
* Patients determined to be suitable for primary simultaneous bilateral TKA based on physical exam and medical history including the following:

  o Osteoarthritis (OA)
* Patient is skeletally mature.
* Patient is willing and able to provide written informed consent.
* Participants must be able to speak and understand Danish
* Patient is willing and able to cooperate in the required post-operative therapy.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent.

Exclusion criteria

* Patients with previous open knee surgery on either knee (i.e., osteotomy, unicompartemental arthroplasty, osteosynthesis)
* Patients with previous major trauma to either knee resulting in deformity og scarring.
* Patients receiving treatment for DVT or PE postoperatively.
* Patients with known allergy to skin adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Wound discharge during stay | 3 days post op
  The wound will be defined as actively oozing, if the standard bandage Mepilex Border Post-op®, is soaked to the border. Bandages soaked to the border will be replaced. Number of replaced bandages for each knee will be recorded.

SECONDARY OUTCOMES:
ASEPSIS score | 3 weeks post op
  Wound healing score

IPD SHARING:
Plan to Share IPD: Undecided